CLINICAL TRIAL: NCT03038594
Title: Growth Hormone Therapy for Muscle Regeneration in Severely Burned Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-0298 / 15-0192; W81XWH-15-1-0143 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2016-05-11; First posted 2017-01-31 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Burns; Growth Hormone Treatment
Keywords: Burns; Growth Hormone; Lean Body Mass; Strength; Exercise Endurance
MeSH Terms: conditions — Burns | interventions — Human Growth Hormone; Growth Hormone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Growth Hormone (Experimental): Daily subcutaneous injections of 0.05 mg/kg/day of Growth Hormone [somatropin, Genotropin, Pfizer, New York, NY] will be administered, from one week prior to discharge until 9 months post-burn.
  Interventions: Drug: Somatropin
- 0.09% saline solution (Placebo Comparator): Daily subcutaneous injections of 0.09% of saline solution will be administered, from one week prior to discharge until 9 months post-burn.
  Interventions: Drug: 0.09% Saline Solution

INTERVENTIONS:
Drug: Somatropin
  Other Names: Genotropin, Growth Hormone (GH)
  Arms: Growth Hormone
Drug: 0.09% Saline Solution
  Other Names: Placebo, Control
  Arms: 0.09% saline solution

SUMMARY:
The investigators have previously demonstrated that burn injury causes severe muscle wasting, weight and height retardation, and systemic protein catabolism in pediatric and adult burned patients. The persistent loss of muscle impairs the quality of life of the burned patients, and it also delays autonomy and reintegration into the community. In 2009, the investigators showed that the daily injection of recombinant human growth hormone (GH) for nine months post discharge significantly increased height and weight, as well as lean body mass, in pediatric burned subjects. Our long-term goal is to improve the quality of life of burn patients by preventing height, weight, and muscle loss that may occur from severe protein catabolism. The objectives of this application are to a) attenuate height and weight in burned patients with the administration of GH, b) prevent or reverse loss of muscle and strength in these patients, and c) collect pilot data about cardiopulmonary parameters, scar assessments, and muscle metabolism. Our central hypothesis is that the administration of GH will restore depleted levels of growth hormone and will lead to prevention of lean body mass loss and bone mineral content, improve rehabilitation, and accelerate reintegration of severely burned patients. The investigators will administer either placebo or GH (daily subcutaneous injections of 0.05 mg/kg/day of GH [somatropin, Genotropin, Pfizer, New York, NY] to adult burn subjects (n=31 per group, 18-85 years, >30% total body surface burns) for nine months beginning one week prior to discharge. Both groups will be studied for a total of two years. The following aims will be tested: 1) determine the effects of GH supplementation on body composition, such as lean body mass loss, muscle strength, and exercise endurance; and 2) assess whether rehabilitation and subsequent reintegration of severely burned patients into society can be accelerated. Investigators will measure changes in lean body mass, muscle strength and exercise endurance during the acute hospital stay, discharge, and long-term follow-up visits (6, 12, 18, and 24 months after burn), as well as secondary endpoints such as cardiopulmonary variables, hypertrophic scar development, quality of life questionnaires, and concentrations of relevant hormones, cytokines, and oxidative stress markers.

DETAILED DESCRIPTION:
Either recombinant human growth hormone (daily subcutaneous injections of 0.05 mg/kg/day of GH at discharge [somatropin, Genotropin, Pfizer, New York, NY]; 0.025 mg/kg/day of GH titrated the week before discharge) or placebo (n=31) will be administered to adult burned subjects (n= 31, 18-85 years) after screening and voluntary consent who have ≥30% TBSA assessed by either the Lund and Browder chart or the 'rule of nines' method during excisional surgery. It will be administered daily for 9 months beginning the week before discharge, and the primary and secondary endpoints will be collected during the acute hospital stay, discharge, and long-term follow-up visits (6, 12, 18, and 24 months after burn injury). Additionally, subjects will be contacted frequently [most likely 1 week, 1 month, and 2 months post discharge by telephone] to ensure that there are no adverse events or concerns with their study drug, as well as visit with them during their clinical visits that address their post-burn needs. All subjects will receive similar standard medical care and treatment from the time of emergency admission until their discharge.

Growth hormone will be used to potentially attenuate losses in height, weight, muscle and bone, reverse the oxidative stress of burn injury and, in the process, decrease the secondary consequences of burn injury, including organ dysfunction. This may improve the quality of life of the burn patient by preventing pathophysiology that may result from muscle and bone loss and may reduce hospital stay. Our research will lay the foundation for the future development of effective, safe, and economic therapeutic interventions to treat burn injury-associated metabolic abnormalities. Also, it will provide the basis for the development of supplemental regulations and pharmacotherapy to treat burn patients with GH. The risks are very reasonable in relation to the anticipated benefits to our subjects because a) GH at a higher dose has been tested in pediatric burned subjects with minor adverse events, and b) the subjects will be monitored consistently.

ELIGIBILITY:
INCLUSION CRITERIA

* 18-85 years old
* Over 30% total body surface area burn
* Provide consent and comprehend English or Spanish

EXCLUSION CRITERIA

* History of AIDS, AIDS-related complex, or HIV
* History of or current hepatitis B or C
* Pregnancy
* History of or Active Malignancy
* Insulin dependent diabetes mellitus type I prior to admission
* Insulin dependent diabetes mellitus type II (up to 12 months prior to admission)
* Other hyperglycemic disorders [not including transient post-burn/trauma hyperglycemia]
* Current oral corticosteroid treatment
* Currently participating in another interventional clinical trial at UTMB

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Lean body mass | At baseline
  Dual-Energy X-ray Absorptiometry (DEXA) measured in grams
Lean body mass | 6 months post burn-injury
  Dual-Energy X-ray Absorptiometry (DEXA) measured in grams
Lean body mass | 12 months post burn-injury
  Dual-Energy X-ray Absorptiometry (DEXA) measured in grams
Lean body mass | 18 months post burn-injury
  Dual-Energy X-ray Absorptiometry (DEXA) measured in grams
Lean body mass | 24 months post burn-injury
  Dual-Energy X-ray Absorptiometry (DEXA) measured in grams

SECONDARY OUTCOMES:
Change in Muscle strength (peak torque) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  resistance testing muscle strength (assessed by Biodex isokinetic dynamometer)
Change in Muscle strength ( total work) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  resistance testing muscle strength (Biodex isokinetic dynamometer)
Change in Muscle strength (average power) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  resistance testing muscle strength (assessed by Biodex isokinetic dynamometer)
Change in Muscle grip strength (maximum power) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  testing muscle strength (assessed by hand dynamometer)
Change in Muscle endurance (maximum power) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  testing muscle endurance (assessed by Bruce treadmill test)
Change in Resting energy expenditure (REE) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Indirect calorimetry
Change in resting heart rate | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  electrocardiogram (EKG) readings
Change in liver size | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Ultrasound readings
Change in cardiac stroke volume | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  echocardiogram readings
Change in cardiac output | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Echocardiogram readings
Change in respiratory quotient | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Indirect calorimetry
Change in Total body fat | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Dual-Energy X-ray Absorptiometry (DEXA)
Change in percentage of total body fat | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Dual-Energy X-ray Absorptiometry (DEXA)
Change in bone mineral content | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Dual-Energy X-ray Absorptiometry (DEXA)
Change in bone mineral density | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Dual-Energy X-ray Absorptiometry (DEXA)
Change in Maximal oxygen consumption | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Six-minute walk test
Change in respiratory fatigue | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Six-minute walk test
Change in leg fatigue | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Six-minute walk test
Change in Muscle protein synthesis rate | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Deuterium water
Hypertrophic scar development | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Vancouver Scar Scale
Change in Forced vital capacity (FVC) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Pulmonary function test
Change in forced expiratory volume in one second (FEV1) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Pulmonary function test
Change in forced expiratory flow rate between 27-75% of the FVC (FEF25-75) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Pulmonary function test
Change in FEV1/FVC ratio expressed as a percentage (FEV1/FVC%) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Pulmonary function test
Change in vital capacity (VC) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Pulmonary function test
Change in total lung capacity (TLC) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Pulmonary function test
Change in residual volume (RV) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Pulmonary function test
Change in functional residual capacity (FRC) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Pulmonary function test
Change in lung diffusion capacity (DLCO) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Pulmonary function test
Change in maximum voluntary ventilation (MVV) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Pulmonary function test
Change in peak expiratory flow (PEF) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Pulmonary function test
Change in Molecular biomarkers of oxidative and nitrosative stress (isoprostanes, asymmetric dimethylarginine) | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Urine analysis
Changes in quality of life | Discharge (usually 30 days post burn) and 6, 12, 18, and 24 months after burn injury
  Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Ludwik K Branski, MD, MMS, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stylianos S, Eichelberger MR. Pediatric trauma. Prevention strategies. Pediatr Clin North Am. 1993 Dec;40(6):1359-68. doi: 10.1016/s0031-3955(16)38666-7. PMID 8255630

DOCUMENTS (1):
  • Informed Consent Form (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT03038594/ICF_001.pdf